CLINICAL TRIAL: NCT03214224
Title: Remote Pulmonary Function Testing in Amyotrophic Lateral Sclerosis (Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Zachary Simmons, Professor of Neurology and Humanities, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006924part1
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Results first posted 2019-04-09 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: ALS
Keywords: Telemedicine; Pulmonary Function Testing; Telehealth

STUDY DESIGN:
Intervention Model Description: A self-controlled validation study of experimental remote PFT assessment vs standard of care (non-randomized)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- remote PFT (rPFT) validation (Experimental): Subjects in this arm perform both standard and remote PFT assessments in order to validate the procedure.
  Interventions: Device: remote pulmonary function testing; Device: standard pulmonary function testing

INTERVENTIONS:
Device: remote pulmonary function testing — Telemedicine delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)
Device: standard pulmonary function testing — Standard clinical delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)

SUMMARY:
The specific objective of this study is to validate the practice of remote pulmonary function testing (rPFT) conducted in the home through the use of connected mobile health devices and the Penn State Hershey ALS Telemanagement program.

DETAILED DESCRIPTION:
The specific objective of this study is to validate the practice of remote pulmonary function testing (rPFT) conducted in the home through the use of connected mobile health devices and the Penn State Hershey ALS Telemanagement program. The central hypothesis is that guided home assessment of respiratory function is a valid method for detecting respiratory insufficiency leading to noninvasive ventilation (NIV) recommendation. This study has the potential to transform the current practice of conducting breathing assessments every three months, resulting in timelier detection of respiratory insufficiency, thereby staining quality of life and lengthening survival. This protocol has the potential to demonstrate telemanagement exceeding the standards of ALS care.

This is a self-controlled study which will enroll 40 patients from the ALS clinic. On the day of their clinical visit, study participants will perform both a standard PFT as well as a simulated rPFT, both generating three valid repetitions of forced vital capacity (FVC) and maximal inspiratory pressure (MIP) procedures. The simulated rPFT will mimic the practice of home telemonitoring by having patients be instructed by a respiratory therapist over the telemanagement portal while in a research room within the ALS clinic. The primary hypothesis is that there is no difference in the results of PFT and rPFT for respiratory assessment of FVC and MIP.

ELIGIBILITY:
Inclusion Criteria:

* Part 1

Patients:

1. Possess a diagnosis of definite, probable, probable laboratory-supported, or possible ALS by revised El Escorial research criteria [Brooks2000].
2. Be 18 years of age or older.
3. Have a caregiver available to participate in the study

Caregivers:

1. Be 18 years of age or older, of either gender.
2. Be able and willing to provide informed consent.

Respiratory Therapist

1. Be a member of the Hershey Medical Center ALS multidisciplinary care team.
2. Be able and willing to provide verbal informed consent after receiving a summary explanation of research (SER).

Part 2 imposes additional inclusion criteria for patients only.

Patients:

4) Symptom onset within the last three years. 5) Have a computer and home internet service sufﬁcient for engaging in telemedicine sessions.

6) Have a second device capable of downloading the spirometer application from an app store (Android- or iOS-based smartphone or tablet).

Exclusion Criteria:

* Exclusion criteria are the same for both parts of the study.

Patients:

1. Use of NIV or diaphragm pacer at time of obtaining informed consent.
2. FVC ≤50% predicted or MIP > -60 cm H2O.
3. ALS Functional Rating Scale (ALSFRS-R) [Cedarbaum1999] score on day of screening of ≥2 on items for speech, swallowing, and salivation. These items are indicators of bulbar dysfunction, which limits the reliability of PFT administration.
4. Cognitive impairment, as judged by the ALS clinic neurologist, that prevents participation in the study.

Caregivers: None

Respiratory Therapists: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hershey Medical Center ALS Clinic, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time to share data with other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 subjects (including 3 patients not completing procedures, 3 controls, and 3 therapists)
Groups:
- Remote PFT (rPFT) Validation: Those in the first part of the study will perform both standard and remote PFT assessments in order to validate the procedure.
Period: Overall Study
Arm/Group | Remote PFT (rPFT) Validation
Started | 49 (Subjects did both standard and remote assessments in the validation study. Total enrollment 49.)
Completed | 40 (3 therapists enrolled. 3 ctrls enrolled (not incl. in analysis). 3 pts enr. but not completed.)
Not Completed | 9
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Practice controls or therapists | 6

BASELINE CHARACTERISTICS:
Population: Only patients who completed validation procedures are included (40 total). Recruitment has not yet begun for the second, randomized phase of the protocol, which involves enrollment into the standard PFT and remote PFT strudy arms.
Groups:
- Remote PFT (rPFT) Validation: Subjects perform both standard and remote PFT assessments in order to validate the procedure.
Arm/Group | Remote PFT (rPFT) Validation
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40
ALS Functional Rating Scale - Revised (ALSFRS-R) [Mean (Standard Deviation); unit: units on a scale] — Scale that measures physical function in bulbar, fine motor, gross motor, and breathing domains. Total score ranges from 0-48. Higher numbers indicate normal function. Lower numbers indicate impaired function.
  units on a scale | 31.3 (7.9)
Time Since Symptom Onset [Mean (Standard Deviation); unit: months] | 59.2 (56.8)
Diagnosis [Count of Participants; unit: Participants]
  ALS | 30
  PLS | 9
  PMA | 1

OUTCOME MEASURES:

1. Primary Outcome: Standard PFT - Forced Vital Capacity
Description: Respiratory therapist will administer three valid maneuvers of forced vital capacity (FVC) The best FVC value is the outcome.
Time Frame: One administration - 10 minutes
Population: 40 patients taking part in validation study
Measure: Mean (Standard Deviation); unit: Percent Predicted FVC
Arm/Group | Remote PFT (rPFT) Validation
Number analyzed (Participants) | 40
Percent Predicted FVC | 72.7 (18.0)

2. Primary Outcome: Standard PFT - Maximal Inspiratory Pressure
Description: Respiratory therapist will administer three valid maneuvers of maximal inspiratory pressure (MIP). The best MIP value is the outcome.
Time Frame: One administration - 10 minutes
Population: 40 patients taking part in validation study
Measure: Mean (Standard Deviation); unit: cm water
Arm/Group | Remote PFT (rPFT) Validation
Number analyzed (Participants) | 40
cm water | -68.7 (26.0)

3. Primary Outcome: Remote PFT - Forced Vital Capacity
Description: Respiratory therapist will use the telehealth interface to guide the patient and caregiver to self-administer three valid FVC maneuvers. The best FVC value is the outcome.
Time Frame: One administration - 10 minutes
Population: 40 patients taking part in validation study
Measure: Mean (Standard Deviation); unit: Percent predicted of FVC
Arm/Group | Remote PFT (rPFT) Validation
Number analyzed (Participants) | 40
Percent predicted of FVC | 79.7 (20.4)

4. Primary Outcome: Remote PFT - Maximal Inspiratory Pressure
Description: Respiratory therapist will use the telehealth interface to guide the patient and caregiver to self-administer three valid MIP maneuvers. The best MIP value is the outcome.
Time Frame: One administration - 10 minutes
Population: 40 patients taking part in validation study
Measure: Mean (Standard Deviation); unit: cm water
Arm/Group | Remote PFT (rPFT) Validation
Number analyzed (Participants) | 40
cm water | -66.2 (28.6)

5. Secondary Outcome: Patient and Caregiver Reported Outcomes
Description: Survey responses from the patient/caregiver pair. Likert-type scales are used to generate subscores pertaining to: General Acceptability, Forced Vital Capacity Acceptability, and Maximal Inspiratory Pressure Acceptability.
  Subscales (evaluated separately):
  General Acceptability [0-5 (worst-best)] Forced Vital Capacity Acceptability [0-5 (worst-best) Maximal Inspiratory Pressure Acceptability [0-5 (worst-best)]
Time Frame: 10 minute survey administered following completion of standard and remote PFT of Part 1
Population: One subject did not complete the survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remote PFT (rPFT) Validation
Number analyzed (Participants) | 39
units on a scale
  General Acceptability | 4.50 (.58)
  Forced Vital Capacity Acceptability | 4.45 (.63)
  Maximal Inspiratory Pressure Acceptability | 4.48 (.59)

6. Secondary Outcome: Therapist Reported Outcomes
Description: Survey responses from the respiratory therapist. Likert-type scales are used to generate subscores pertaining to: General Acceptability, Forced Vital Capacity Acceptability, and Maximal Inspiratory Pressure Acceptability.
  Subscales (evaluated separately):
  General Acceptability [0-5 (worst-best)] Forced Vital Capacity Acceptability [0-5 (worst-best) Maximal Inspiratory Pressure Acceptability [0-5 (worst-best)]
Time Frame: 10 minute survey administered following completion of standard and remote PFT of Part 1
Population: There were three therapists who produced 35 separate survey responses. Responses from 5 patient interactions were not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remote PFT (rPFT) Validation
Number analyzed (Participants) | 35
units on a scale
  General Acceptability | 4.16 (.50)
  Forced Vital Capacity Acceptability | 3.75 (.63)
  Maximal Inspiratory Pressure Acceptability | 4.04 (.44)

ADVERSE EVENTS:
Time Frame: For the validation study, adverse event data was collected over the period of the procedures, approximately 20 minutes.
Arm/Group | Remote PFT (rPFT) Validation
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03214224/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT03214224/ICF_001.pdf